CLINICAL TRIAL: NCT01607970
Title: Double-blind, Placebo-controlled, Randomized Study: Oxytocin Modulation of Startle Reactivity to Social Stimuli and Moral Decision Making
Brief Title: Oxytocin Modulation of Startle Reactivity to Social Stimuli and Moral Decision Making
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Rene Hurlemann, MSc MD PhD, University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: OXT-168/11
Record Dates: First submitted 2012-05-23; First posted 2012-05-30 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Healthy Male Volunteers
Keywords: Oxytocin; Startle; moral dilemma; oxytocin receptor gene
MeSH Terms: interventions — Oxytocin; lactitol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin (Experimental): 24 IU Oxytocin, intranasal application 45 min prior to the experiment
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): intranasal application, sodium chloride solution, 3 puffs per nostril
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin: 24 IU; 3 puffs per nostril, each with 4 IU OXT
  Other Names: Oxytocin: Syntocinon-Spray, Novartis

SUMMARY:
The purpose of this study is to determine whether oxytocin affects the modulation of startle reactivity by aversive social stimuli and to investigate the oxytocin effect on moral judgements. Furthermore the investigators explore the effects of oxytocin receptor (OXTR) polymorphisms on behavioral responses to social stimuli.

DETAILED DESCRIPTION:
The neuropeptide oxytocin (OXT) can enhance the impact of positive social cues but may reduce that of negative ones, although it is unclear whether the latter causes blunted emotional responses. After OXT or placebo application participants are exposed to acoustic startle probes presented alone and during viewing of 60 color pictures mostly selected from the 'International Affective Picture System'. The paradigm featured 20 negative (mostly threatening), 20 neutral, and 20 positive pictures, presented for 5 s each. In the other part of the experiment, after intranasal OXT or placebo application participants respond to 60 moral dilemmas.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers

Exclusion Criteria:

* Current or past psychiatric disease
* Current or past physical illness
* Psychoactive medication
* Tobacco smokers

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
baseline startle magnitude and affective modulation of the startle magnitude after oxytocin and placebo administration | 24 Months
  The experimental tasks started 45 min after intranasal OXT/PLC administration. The STARTLE-paradigm features 20 negative (mostly threatening), 20 neutral, and 20 positive pictures, presented for 5 s each. The startle stimulus consists of a single 50-ms burst of white noise (100 dB) with nearly instantaneous rise and was delivered binaurally via headphones during 60% of the pictures (i.e. 12 from each category) at 2 - 4 s after picture onset. We examined the baseline startle magnitude as well as the affective modulation of the startle magnitude.

SECONDARY OUTCOMES:
moral decision making after oxytocin and placebo administration | 24 months
  The experimental tasks started 45 min after OXT/PLC administration. The moral dilemmas performed in the present study were identical to those published previously by Greene et al.(2001).
oxytocin receptor (OXTR) polymorphism and correlation with social behavior | 24 months
  OXTR genotyping, social behavior testing

CONTACTS AND LOCATIONS:
Overall Officials: Rene Hurlemann, MSc MD PhD, Principal Investigator — Department of Psychiatry, University of Bonn, Germany
Locations (1):
- Department of Psychiatry, University of Bonn, Bonn, Germany

REFERENCES:
- See also: Click here for more information about the NEMO research group — http://renehurlemann.squarespace.com/welcome/